CLINICAL TRIAL: NCT05029609
Title: A Phase 1b, Double-Blind, Randomized, Placebo Controlled, Multiple Ascending Dose Study of the Safety, Tolerability and Immune Effects of the Intranasal Anti-CD3 Monoclonal Antibody Foralumab in Primary and Secondary Progressive MS
Brief Title: Phase 1b Multiple Ascending Dose Study of Foralumab in Primary and Secondary Progressive MS
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawn due to business reasons
Sponsor: Tiziana Life Sciences LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TILS-015
Record Dates: First submitted 2021-08-27; First posted 2021-08-31 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Primary Progressive Multiple Sclerosis; Secondary Progressive Multiple Sclerosis; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: This is a Phase 1b double blind, randomized, placebo controlled, dose escalating study evaluating multiple doses of Foralumab via intranasal administration for 14 days in patients with MS.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A (Other): Group A will receive nasal Foralumab Dose 1 daily for 14 days (n=9) or placebo (n=3)
  Interventions: Drug: Intranasal Foralumab Solution; Drug: Placebo
- Group B (Other): Group B will receive nasal Foralumab Dose 2 tiw for 14 days (n=9) or placebo (n=3)
  Interventions: Drug: Intranasal Foralumab Solution; Drug: Placebo
- Group C (Other): Group C will receive nasal Foralumab Dose 3 daily for 14 days (n=9) or placebo (n=3)
  Interventions: Drug: Intranasal Foralumab Solution; Drug: Placebo
- Group D (Other): Group D will receive nasal Foralumab Dose 4 daily for 14 days (n=9) or placebo (n=3)
  Interventions: Drug: Intranasal Foralumab Solution; Drug: Placebo

INTERVENTIONS:
Drug: Intranasal Foralumab Solution — The Aptar Unidose device will be used to deliver foralumab nasal solution intranasally. Foralumab nasal solution is prepackaged in a Type 1 glass vial inside the Unidose device.
Drug: Placebo — The placebo nasal solution is the acetate buffer vehicle used for foralumab nasal solution. It will be handled in a manner identical to active drug.

SUMMARY:
The primary objective is to establish the safety of administration of intranasal Foralumab in non-active primary and secondary progressive Multiple Sclerosis (MS) patients in a multiple ascending dose format in escalating doses for 14 consecutive days.

DETAILED DESCRIPTION:
This is a Phase 1b double blind, randomized, placebo controlled, dose escalating study evaluating multiple doses of Foralumab via intranasal administration for 14 days in patients with MS.

Up to 55 untreated primary and secondary progressive MS patients will be enrolled, to obtain a total of 48 completed subjects (9 active, 3 placebos per group), allowing for dropouts.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of MS (according to the 2010 McDonald criteria).
2. Age 25-70 years.
3. Clinical diagnosis of non-active primary and secondary MS
4. MRI imaging consistent with a diagnosis of MS at any time point.
5. Score on the Expanded Disability Status Scale (EDSS) of 2.5-6.5
6. Adequate hematologic parameters without ongoing transfusion support:

   * Hemoglobin (Hb) ≥ 9 g/dL
   * Platelets ≥ 100 x 109 cells/L
7. Creatinine ≤ 1.5 x the upper limit of normal (ULN), or calculated creatinine clearance

   ≥ 60 mL/minute x 1.73 m2 per the Cockcroft-Gault formula
8. Total bilirubin ≤ 2 times the upper limit of normal (ULN) unless due to Gilbert's disease
9. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN, or < 5 times ULN for patients with liver metastases
10. QT interval corrected for rate (QTcF) ≤ 470 msec for women and ≤ 450 msec for men on the ECG obtained at Screening
11. Negative serum pregnancy test within 14 days prior to the first dose of study therapy for women of child-bearing potential (WCBP)

13. Ability to provide written informed consent.

Exclusion Criteria:

1. Corticosteroid use (oral or intravenous) within the last 30 days.
2. Current use or use in the prior 6 months of MS immunotherapy, interferon, glatiramer acetate, fingolimod, siponimod, dimethyl fumarate or natalizumab or any other chronic immunosuppressive medication
3. Inability to tolerate intranasally administered medications
4. Nasal corticosteroids, nasal antihistamines, nasal flu dosing within the past 30 days.
5. Chronic rhinitis, deviated septum, nasal polyps, history of sinusitis treated within the past 12 months.
6. Active COVID-19 disease; according to FDA guidelines
7. Female patient who is pregnant, lactating, breastfeeding, or planning on becoming pregnant during study.
8. Female patients of childbearing age will undergo a pregnancy test and be excluded from the study if positive.
9. Active malignancy within 5 years.
10. Inflammatory bowel disease, rheumatoid arthritis, systemic lupus erythematosus, asthma, or type 1 diabetes
11. Neutropenia (<500 neutrophils/mL) or other severe immunosuppression
12. Unable or unwilling to comply with protocol requirements.
13. Patients with a history of gadolinium allergy.
14. Screening labs outside of the normal range; EBV IgM positive subjects with clinical signs will not receive study drug.
15. Serious cardiac condition within the last 6 months, such as uncontrolled arrhythmia, myocardial infarction, unstable angina or heart disease defined by the New York Heart Association (NYHA) Class III or Class IV (See Appendix B) or hereditary long QT syndrome
16. Concomitant medication(s) that may cause QTc prolongation or induce Torsades de Pointes, except for antimicrobials that are used as standard of care to prevent or treat infections and other such drugs that are considered by the Investigator to be essential for patient care
17. Known positive for human immunodeficiency virus (HIV), hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV)
18. Any other medical intervention or other condition which, in the opinion of the Principal Investigator, could compromise adherence to study requirements or confound the interpretation of study results

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
To establish the safety of intranasal foralumab in non-active primary and secondary progressive MS in escalating doses for 14 consecutive days | 14 days
  Analyses through review of adverse events categorized and graded via CTCAE.

SECONDARY OUTCOMES:
Change in Expanded Disability Status Scale (EDSS) at Day 45 | 45 days
  The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist. EDSS steps 1.0 to 4.5 refer to people with MS who are able to walk without any aid and is based on measures of impairment in eight functional systems. Lower score indicates that the subject is doing better.

IPD SHARING:
Plan to Share IPD: No